CLINICAL TRIAL: NCT04762797
Title: Management Strategy of Polypoid Lesions of the Gallbladder: a Single-center Retrospective Cohort Study
Brief Title: Management Strategy of Polypoid Lesions of the Gallbladder
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCHTF3
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2015-01

CONDITIONS: Polyp Gallbladder
Keywords: gallbladder polyp; laparoscopic cholecystectomy; polypectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-neoplastic group: Gallbladder polyps with pathological diagnosis of cholesterol polyps or inflammatory polyps are classified into "Non-neoplastic group".
  Interventions: Other: Non
- Neoplastic group: Gallbladder polyps pathologically diagnosed as adenocarcinoma, adenoma, adenomyosis, or other malignancies are classified into "Neoplastic group".
  Interventions: Other: Non

INTERVENTIONS:
Other: Non — This is a retrospective study, without intervention.

SUMMARY:
We retrospectively review a single-center cohort of gallbladder polyps from January 2015 to May 2020. Univariate and multivariable analyses were performed to extract potential risky factors of neoplastic polyps. Also, a comparison was conducted between laparoscopic cholecystectomy (LC) and laparoscopic polypectomy (LP) to explore factors affecting surgeons' decision on LC or LP.

ELIGIBILITY:
Inclusion Criteria:

Surgical indications for LC included polyp diameter over 10 millimeters, or polyps accompanied by GB stones, or consideration of neoplastic polyps. Surgical indications for GB-preserving surgery included GB with normal emptying function and polyp diameter smaller than 10 millimeters, or consideration of benign non-neoplastic polyps, or asymptomatic polyps.

Exclusion Criteria:

Those do not fit for laparoscopic surgery.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: surgical candidates of laparoscopic cholecystectomy or laparoscopic polypectomy.
Sampling Method: Non-Probability Sample
Enrollment: 672 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Pathological diagnosis of polyps | Up to two weeks after surgery
  Pathological diagnosis of polyps

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Qu, Doctor, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided